CLINICAL TRIAL: NCT05814783
Title: A Clinician Training Program to Integrate Digital Cognitive Behavior Therapy for Insomnia Into Routine Psychotherapy
Brief Title: Clinician Training Program to Integrate Digital CBTI Into Routine Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Sleep Research Society Foundation (Unknown)
Responsible Party: Principal Investigator, Nicole Gumport, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68391
Record Dates: First submitted 2023-03-01; First posted 2023-04-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Integrated digital CBTI (Experimental): Therapists will be trained to integrate digital CBTI alongside routine psychotherapy. Patients will receive integrated digital CBTI
  Interventions: Behavioral: supported digital CBTI; Device: digital CBTI

INTERVENTIONS:
Behavioral: supported digital CBTI — in session support for adherence to and engagement with digital CBTI
Device: digital CBTI — CBTI app

SUMMARY:
The goal of this study is to pilot test and refine a training program for licensed therapists to promote the integration of digital cognitive behavior therapy for insomnia (dCBTi) into their routine mental health care services.

ELIGIBILITY:
Therapist Criteria:

Inclusion Criteria:

* Licensed mental health clinicians
* Have a clinical care model that includes seeing patients weekly or biweekly
* Provide therapy in English
* Treat patients with depression and/or anxiety
* Can identify 1-2 patients who are willing to consent to be training cases.

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Patient Criteria:

Inclusion Criteria:

* Aged 18+ years old
* Receive weekly or biweekly therapy from participating study therapist
* Identify improving sleep as a goal for treatment and experience insomnia (Insomnia Severity Index score greater than or equal to 10)
* Have daily access to a smartphone, tablet, or computer
* Can read, write, and speak in English

Exclusion Criteria:

* Conditions known to make study treatment less effective (e.g., current chronic medication use known to interfere with sleep, alcohol or substance use disorder, thought disorder)
* Conditions for which dCBTi is a safety risk (e.g., bipolar disorder, excessive daytime sleepiness)
* Current psychotherapy for insomnia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Pre-treatment and immediately post-treatment (treatment phase is 12 weeks)
  Validated questionnaire; total score range between 0 and 28, with higher numbers representing greater insomnia severity, patient outcome.
Change in Knowledge of Supporting Integrated dCBTi | Pre-training (at the start of the one day training) and immediately post-training (at the end of the one day training)
  Therapist outcome assessing knowledge gained during training program measured via a study-specific questionnaire on which higher scores indicating more knowledge

SECONDARY OUTCOMES:
Time spent supporting dCBTi | Through study duration, usually 3 months
  From a structured post-session note completed by the therapist, therapist-reported how much time spent devoted to supporting dCBTI

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Gumport, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No